CLINICAL TRIAL: NCT05642156
Title: Hemodynamics in Chronic Hemodialysis Patients Undergoing Isolated Ultrafiltration Compared to Conventional Hemodialysis
Acronym: ISO-UF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ISO-UF
Record Dates: First submitted 2022-11-17; First posted 2022-12-08 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-03

CONDITIONS: End Stage Kidney Disease
Keywords: hemodialysis; ultrafiltration
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequential HD - Conventional HD (Active Comparator): In sequence A patients will be treated with sequential HD first, for a total of 8 session and then switched to a conventional HD schedule for another 8 sessions.
  Interventions: Procedure: isolated Ultrafiltration (iso-UF)
- Conventional HD - Sequential HD (Active Comparator): In sequence A patients will be treated with conventional HD first, for a total of 8 session and then switched to a sequential HD schedule for another 8 sessions.
  Interventions: Procedure: isolated Ultrafiltration (iso-UF)

INTERVENTIONS:
Procedure: isolated Ultrafiltration (iso-UF) — isolated Ultrafiltration

SUMMARY:
Patients treated with hemodialysis (HD) bear increased risk of cardiovascular events, which results in high morbidity and mortality among this cohort of patients. Intradialytic hypotension (IDH), which is an independent risk factor for mortality, occurs in up to 20% of hemodialysis session and may lead to myocardial stunning and cerebral ischemia resulting in increased white matter lesions, gastrointestinal ischemia and shunt vessel thrombosis. Due to the deleterious effects of IDH during HD, preventive measurements such as limiting interdialytic weight gain are recommended, but frequently fluid and salt restriction are not adhered to, thus increasing dialysis time or frequency of treatments is a common strategy in those patients.

DETAILED DESCRIPTION:
A KDIGO (Kidney Disease: Improving Global Outcomes) controversies conference suggested that isolated ultrafiltration (iso-UF) may provide a benefit in hemodynamic stability, but whether this translates into benefits in hard outcomes is unclear and requires further research. So called-sequential dialysis, that is, isolated ultrafiltration followed by HD is commonly recommended, but evidence is very limited and mainly based on small older studies.

In conclusion, the supposed benefit for intradialytic hemodynamic stability attributed to isolated ultrafiltration compared to hemodialysis seems to be due to less pronounced changes in vascular resistance, but the reason for this discrepancy is unclear. Thus far, recommendations for using iso-UF to improve hemodynamic stability are mainly based on old studies which may not be applicable to modern technique used nowadays. Furthermore, there is no standardized approach on how to use isolated ultrafiltration, with neither a time period nor ultrafiltration rate recommended by the guidelines.

In this study, the investigators try to assess changes in peripheral resistance, osmolality, cardiac output, and cardiac power index and try to establish exploratory correlations to IDH episodes. Furthermore, the investigators want to assess the impact on dialysis quality by reduced time on dialysis.

ELIGIBILITY:
Inclusion Criteria:

* Written consent of the participant after being informed
* At least 18 years of age
* End stage kidney disease patient undergoing hemodialysis
* Dry weight stable for a minimum of one month
* Interdialytic weight gain of >2 liters in the short interdialytic interval

Exclusion Criteria:

* No informed consent was obtained
* Patients with a pacemaker or implanted medical device that prevents compliance with study regulations
* Patients treated with hemodiafiltration
* Patients treated with medium cut-off membranes (Theranova, Baxter)
* Patients with recurrent severe hyperkalemia after the short interdialytic interval (K+ concentration > 6.0 mmol/L, requiring more than 2 hours of dialysis to ameliorate the post-dialytic shift from other compartments.
* Women of childbearing age not using contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2022-11-02 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Total peripheral resistance index (TPRI) | up to 8 weeks
  Absolute change of TPRI (expressed as dyn*sec/cm*m2) in each individual session from baseline to the nadir.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Graz, Graz, Austria

IPD SHARING:
Plan to Share IPD: No